CLINICAL TRIAL: NCT01730690
Title: Bacterial Meningitis in Adults: Analysis of the Determinants of Mortality and Neurosensory Sequelae
Acronym: COMBAT
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: CRC11040; NI11046 (Other: APHP)
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Meningitis, Bacterial
Keywords: Bacterial meningitis in adults; determinants of in-hospital mortality
MeSH Terms: conditions — Meningitis, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Major changes in the epidemiological characteristics of bacterial meningitis have been observed as a result of changes in behaviour, human interventions (use of antibiotics, prophylactic vaccinations), as well as poorly elucidated mechanisms responsible for epidemic outbreaks.

The objective of this study is to identify the determinants of in-hospital mortality of bacterial meningitis in adults.

Hypothesis : the standardized data collection concerning cases of bacterial meningitis in adults with telephone follow-up would allow analysis of the determinants of mortality and neurosensory sequelae, description of the psychosocial impact and proposal of new treatment strategies.

DETAILED DESCRIPTION:
Introduction: Bacterial meningitis is a rare (about 1,200 cases per year in France, 50% occurring in adults) and serious disease (20% mortality during the acute phase; neurosensory sequelae in 30% of survivors). Major changes in the epidemiological characteristics of bacterial meningitis have been observed as a result of changes in behaviour, human interventions (use of antibiotics, prophylactic vaccinations), as well as poorly elucidated mechanisms responsible for epidemic outbreaks. No standardized clinical, microbiological and prognostic data collection concerning bacterial meningitis in adults is available in France.

Hypothesis: Standardized data collection concerning cases of bacterial meningitis in adults with telephone follow-up would allow analysis of the determinants of mortality and neurosensory sequelae, description of the psychosocial impact and proposal of new treatment strategies.

Primary objective: To identify the determinants of in-hospital mortality of bacterial meningitis in adults.

Secondary objectives: To describe the epidemiological characteristics of community-acquired bacterial meningitis in adults, changes in these characteristics and their relations with the vaccine status of the affected adult and his/her family; to characterize clinical and microbiological failures and their determinants (pharmacological, microbiological, immunological, etc.); to analyse the determinants of neurosensory sequelae and failure to return to work after 1 month, 6 months and 12 months.

Primary endpoint: In-hospital mortality (D30). Secondary endpoints: History including vaccination of the case and the family, clinical, microbiological (species, susceptibility, virulence factors, cerebrospinal fluid CSF) culture on D0 and H48), imaging characteristics; treatments, CSF antibiotic concentrations, neurological sequelae (modified Rankin, Glasgow Outcome Scale, IQCODE) at M1, M6 an M12, quality of life test SF12, WHO QoL, CESD) at M1, M6, M12, hearing loss (audiometric tests, hereditary hearing impairment (HHI), telephone speech test in noise) at M1, M6, M12.

Methodology, study design: National observational cohort study with comprehensive recruitment in participating centres.

Legal classification of the project: Epidemiological study. Number of subjects required: The inclusion of 150 cases of meningitis per year would allow the collection of about 450 cases over a period of 3 years. For a mortality rate of 20%, we would be able to estimate this percentage with a confidence interval of ± 3.7% (95% confidence interval: 16.3-23.7). With 90 deaths, a power of 80% and a level of significance of 5% (two-tailed), this sample size would demonstrate relative risks of 1.8 for a prevalence of the risk factor of 25% and 2.6 for a prevalence of the risk factor of 10%.

Inclusion criteria: Adult with community-acquired bacterial meningitis defined by the presence of at least one of the following criteria: 1/ Positive CSF culture and/or positive soluble antigen in CSF with or without cell reaction; 2/ Positive PCR in CSF; 3/ Purpura fulminant (with or without positive CSF culture); Positive polymerase chain reaction (PCR) in blood and/or positive blood culture AND CSF cell reaction.

Non inclusion criteria: Age less than 18 years old or refusal to participate. Inclusion period: 3 years. Duration of participation for one patient: 12 months. Number of participating centers: Constitution in participating centers of a dual investigator team comprising a clinician (infectious diseases physician, intensive care physician, or neurologist) and a microbiologist (participating in the national network of "OBSERVATOIRES REGIONAUX DU PNEUMOCOQUE" [Regional Pneumococcal Observatories]). Declaration by the microbiologist to the data management centre. On-site validation of cases by the dual investigator team and then by a national multidisciplinary validation unit.

Mean number of inclusions per month and per centre: 0.5

ELIGIBILITY:
Inclusion Criteria:

* Positive CSF culture and/or positive soluble antigens in CSF with or without a cell reaction
* Positive PCR in CSF
* Purpura fulminant (with or without positive CSF culture)
* Positive PCR in blood and/or positive blood culture AND CSF cell reaction.

Exclusion Criteria:

* Age less than 18 years old
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with bacterial meningitis adults
Sampling Method: Non-Probability Sample
Enrollment: 527 (Actual)
Dates: Start 2013-03; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | 30 days
  mortality in hospital at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Xavier duval, Principal Investigator — APHP
Locations (1):
- Assistance Publique des Hôpitaux de Paris, Paris, France

REFERENCES:
- [Derived] Van RN, Tubiana S, De Broucker T, Cedric J, Roy C, Meyohas MC, Prazuck T, Chirouze C, Hoen B, Duval X, Revest M; COMBAT study group. Persistent headaches one year after bacterial meningitis: prevalence, determinants and impact on quality of life. Eur J Clin Microbiol Infect Dis. 2023 Dec;42(12):1459-1467. doi: 10.1007/s10096-023-04673-y. Epub 2023 Oct 23. PMID 37867184
- [Derived] Della Vecchia C, Ebah JV, Tubiana S, Guimard T, Piroth L, Jaffuel S, Gorenne I, Mourvillier B, Hoen B, Duval X, Preau M. Mid-term health-related quality of life in community-acquired bacterial meningitis survivors; the COMBAT study. PLoS One. 2023 Mar 23;18(3):e0281544. doi: 10.1371/journal.pone.0281544. eCollection 2023. PMID 36952472
- [Derived] Akroum S, Tubiana S, de Broucker T, Dournon N, Varon E, Ploy MC, Mourvillier B, Oziol E, Lacassin F, Laurichesse H, Hoen B, Duval X, Burdet C; and the COMBAT study group. Long-term neuro-functional disability in adult patients with community-acquired bacterial meningitis. Infection. 2022 Oct;50(5):1363-1372. doi: 10.1007/s15010-022-01855-2. Epub 2022 Jun 3. PMID 35657529
- [Derived] Duval X, Taha MK, Lamaury I, Escaut L, Gueit I, Manchon P, Tubiana S, Hoen B; COMBAT study group. One-Year Sequelae and Quality of Life in Adults with Meningococcal Meningitis: Lessons from the COMBAT Multicentre Prospective Study. Adv Ther. 2022 Jun;39(6):3031-3041. doi: 10.1007/s12325-022-02149-7. Epub 2022 Apr 28. PMID 35484469
- [Derived] Benadji A, Duval X, Danis K, Hoen B, Page B, Beraud G, Vernet-Garnier V, Strady C, Brieu N, Maulin L, Roy C, Ploy MC, Gaillat J, Varon E, Tubiana S; COMBAT Study Group; SIIP Study Group. Relationship between serotypes, disease characteristics and 30-day mortality in adults with invasive pneumococcal disease. Infection. 2022 Feb;50(1):223-233. doi: 10.1007/s15010-021-01688-5. Epub 2021 Sep 1. PMID 34468953
- [Derived] Tubiana S, Varon E, Biron C, Ploy MC, Mourvillier B, Taha MK, Revest M, Poyart C, Martin-Blondel G, Lecuit M, Cua E, Pasquet B, Preau M, Hoen B, Duval X; COMBAT study group. Community-acquired bacterial meningitis in adults: in-hospital prognosis, long-term disability and determinants of outcome in a multicentre prospective cohort. Clin Microbiol Infect. 2020 Sep;26(9):1192-1200. doi: 10.1016/j.cmi.2019.12.020. Epub 2020 Jan 10. PMID 31927117